CLINICAL TRIAL: NCT06957002
Title: Bosentan in the Treatment of Giant Cell Arteritis. Multicenter, Randomized, Controlled, Superiority Phase II Trial Comparing a Combination of Bosentan and Glucocorticoids Versus Glucocorticoids Alone in the Treatment of Patients With GCA
Brief Title: Bosentan in the Treatment of Giant Cell Arteritis
Acronym: BOSICART
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P200041; 2024-517030-17 (EudraCT Number)
Record Dates: First submitted 2025-03-24; First posted 2025-05-04 (Actual); Last update posted 2025-05-14 (Actual); Status verified 2025-05

CONDITIONS: Giant Cell Arteritis (GCA)
Keywords: Giant Cell Arteritis; Bosentan
MeSH Terms: conditions — Giant Cell Arteritis | interventions — Bosentan; Glucocorticoids

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Bosentan + Glucocorticoids (Experimental): Bosentan : 62.5 mg bid for 4 weeks and 125 mg bid during 9 additional weeks Glucocorticoids : prespecified GC tapering schedule
  Interventions: Drug: Bosentan
- Glucocorticoids (Other): prespecified GC tapering schedule
  Interventions: Drug: Glucocorticoids

INTERVENTIONS:
Drug: Bosentan — Bosentan : 62.5 mg twice a day for 4 weeks and 125 mg twice a day during 9 weeks (treatment length 3 months)
  Arms: Bosentan + Glucocorticoids
Drug: Glucocorticoids — prespecified GC tapering schedule
  Arms: Glucocorticoids

SUMMARY:
The purpose of this study is to determine whether a treatment with 3 months of bosentan associated to standard therapy might be superior to glucocorticoids alone in term of failure free survival at 12 months

DETAILED DESCRIPTION:
Giant cell arteritis (GCA) is the most common vasculitis in individuals over the age of 50. It is characterized by inflammation of large vessels, including the aorta and its main branches. Patients experience headaches, scalp tenderness, joint pain, and general symptoms such as weight loss, fatigue, and fever. More rarely, unilateral or bilateral visual acuity is impaired. At the biological level, an increase in inflammatory markers, such as C-reactive protein (CRP), is observed.

Glucocorticoids (GCs) are the cornerstone of GCA treatment and are usually administered for 12 to 18 months to prevent relapse, sometimes longer. However, most patients develop significant adverse effects associated with GCs, including hypertension, arterial disease, diabetes, osteoporosis, and infections. As a result, various strategies targeting the inflammatory process have been developed to reduce GC use. For example, methotrexate has been shown to be a modestly effective GC-sparing treatment. A 12-month course of tocilizumab (TCZ), an interleukin-6 (IL-6) receptor antagonist, has also been shown to induce and maintain remission of GCA, with a significant GC-sparing effect. However, only 45% of patients remained in long-term remission after discontinuing tocilizumab.

In patients with GCA, in addition to lymphocyte (white blood cell) activation, the investigator observed increased proliferative properties of vascular smooth muscle cells (VSMCs), obtained from temporal artery biopsies at the time of diagnosis. This proliferation and migration of VSMCs are promoted by endothelin-1 (ET-1), a molecule expressed in the walls of diseased arteries. Thus, ET-1 contributes to vessel lumen narrowing and complete obstruction. It was found that plasma ET-1 concentrations were higher in patients with visual ischemic complications. Additionally, an association was found between endothelin expression in temporal artery biopsies at baseline and therapeutic response at month six.

Bosentan has been marketed since 2002 for the management of patients with pulmonary arterial hypertension. This vasodilating drug is an endothelin (ET-1) receptor antagonist.

The investigator hypothesize that a 3-month course of treatment with bosentan, an endothelin receptor antagonist, combined with standard therapy, could be more effective than glucocorticoids (GCs) alone, reducing the risk of relapse and the current adverse effects, thereby improving relapse-free survival at 12 months.

ELIGIBILITY:
* Inclusion Criteria :
* Patients having given their written informed consent prior to participation in the study
* Patients affiliated with social security or CMU (profit or being entitled)
* Diagnosis of GCA, as defined by the revised GCA diagnosis criteria. Patients must satisfy criteria 1-2-3 and 4 (irrespective of time):

  * Age ≥50 years at disease onset
  * History of erythrocyte sedimentation rate (ESR) ≥ 50 mm/h or CRP ≥ 20 mg/L (not mandatory if TAB is positive: see below)
  * At least one of the following:
* unequivocal cranial symptoms of GCA (new onset headache, scalp tenderness, jaw claudication, temporal artery abnormality, ischemia-related vision loss)
* unequivocal symptoms of polymyalgia rheumatica (PMR)

  * At least one of the following:
* Temporal artery biopsy (TAB) compatible with the diagnosis of GCA (non-necrotizing vasculitis with a predominance of mononuclear cell infiltration or granulomatous inflammation, usually with multinucleated giant cells)
* Evidence of large vessel vasculitis:

  * angio-CT or angio-MRI: thickened and/or contrast-enhanced arteries especially aorta (≥2mm) and epiaortic arteries (≥1mm) and contrast enhanced arteries in T1-weighted sequences
  * or PET scan: ≥ grade 2 (from 0 to 3) tracer uptake on large arteries
* At least a sign of active GCA within the 2 weeks prior to randomisation. Active GCA is defined by ESR ≥30 mm/h or CRP ≥10 mg/L and at least one of the following:
* unequivocal cranial symptoms of GCA (new onset localized headache, scalp or temporal artery tenderness, ischemia-related vision loss, or otherwise unexplained mouth or jaw pain upon mastication)
* unequivocal symptoms of PMR, defined as shoulder and/or hip girdle pain associated with inflammatory stiffness
* other features judged by the clinical investigator to be consistent with GCA or PMR flares
* Menopausal women (no gynaecological cycle over the past two years), or women who had a gynaecological cycle within previous 24 months (non-menopausal women) only if they have (1) an effective non hormonal contraceptive method throughout study and (2) a negative urinary beta-hCG test at inclusion.

Exclusion Criteria:

* Patients under maintenance of justice, wardship or legal guardianship
* Patient unable to give written informed consent prior to participation in the study
* Patients included in other investigational therapeutic study within the previous 3 months
* Patients suspected not to be observant to the proposed treatments
* Weight <40 Kg or > 100 Kg
* Moderate to severe hepatic impairment, i.e., Child-Pugh class B or C. History of chronic alcohol abuse (consumption > 20 g/day)
* Severe chronic heart failure or severe systolic dysfunction
* Recent (< 3 months) or incoming surgery requiring a general anaesthesia
* History of stem cell or organ transplantation (except corneas if performed more than 3 months prior inclusion)
* Hypersensitivity to bosentan or one of its excipients
* Prior treatment with any of the following:

  * Tocilizumab or methotrexate or secukinumab within 12 weeks preceding inclusion
  * Cell-depleting agents (i.e., anti-CD20)
  * Alkylating agents including cyclophosphamide
  * Hydroxychloroquine, cyclosporine A, dapsone, azathioprine, mycophenolate mofetil or janus kinase inhibitors within 4 weeks preceding inclusion
  * Tumor necrosis factor inhibitors within 8 weeks preceding inclusion
  * Anakinra within 1 week preceding inclusion
* Ongoing treatment with glibenclamide, fluconazole and rifampicin. Concomitant administration of both a CYP3A4 inhibitor or a CYP2C9 inhibitor
* Long-course systemic glucocorticoid therapy for other conditions than GCA or PMR
* Laboratory abnormalities: AST or ALT >3 x upper limit of normal (ULN)
* Infections:

  * Active hepatitis B or C
  * HIV infection

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-09 (Estimated); Primary Completion 2029-09 (Estimated); Study Completion 2029-09 (Estimated)

PRIMARY OUTCOMES:
Failure free survival at Week 52 | 12 months ( Week 52)
  A failure is defined by the occurrence of a relapse or the impossibility to decrease Glucocorticoids according to the predefined scheduled Glucocorticoids scheme.

SECONDARY OUTCOMES:
Proportion of new ischemic event | 12 months (Week 52)
Proportion of patients in remission without prednisone | 12 months (Week 52)
  Proportion of patients in remission without prednisone
Proportion of patients in remission with prednisone ≤5 mg/day | 12 months (Week 52)
Cumulative dose of prednisone | 12 months (Week 52)
Proportion of patient in remission | 2 years
  Proportion of patient in remission
Proportion of patients relapsing | year 1 to year 2
  Proportion of patients relapsing
Proportion of patients receiving Glucocorticoids | 2 years
Quality of life measured by the "Health Assessment Questionnaire" (HAQ) | at Week 26 and Week 52
  HAQ (Health Assessment Questionnaire) is a functional disability tool specific to rheumatoid arthritis. The assessment covers the past week and 8 domains of physical activity. For each area of activity, 2 to 3 items are described. Each item can be modified with aids. Only items with a specified response or aid are taken into account. Scores range from 0 (no impact) to 3 (maximum impact).
Quality of life measured by the "Short Form 36 Questionnaire" (SF36) | at Week 26 and Week 52
  To score the SF-36, scales are standardized with a scoring algorithm or by the SF-36 (v2) scoring software to obtain a score ranging from 0 to 100. Higher scores indicate better health status, and a mean score of 50 has been articulated as a normative value for all scales
Frequency and type of side effects | within 1 year after inclusion
  Frequency and type of side effects
Exploratory criteria | At the beginning of the study and in both groups at Week 13 and Week 52
  Compare the remodeling cytokines (pentraxin 3, osteoprotegerin, osteopontin, osteocalcin, thrombomodulin, HGF, endothelin, IL-6, TGF-β MMP-3)

CONTACTS AND LOCATIONS:
Overall Officials: Luc MOUTHON, Pr, Study Director — Hôpital Cochin, Department of Internal Medicine - 75014, Paris
Locations (1):
- Unité de Recherche Clinique, Entrepôts de données et Pharmacologie GHU Paris Centre, Paris, France

IPD SHARING:
Plan to Share IPD: No